CLINICAL TRIAL: NCT05231863
Title: Tyrosine Kinase Inhibitors (TKIs) Based Therapy in Trastuzumab Emtansine (T-DM1) Resistant HER2-positive Metastatic Breast Cancer: A Real-world Study
Brief Title: Tyrosine Kinase Inhibitors (TKIs) in Trastuzumab Emtansine (T-DM1) Resistant HER2-positive Metastatic Breast Cancer: A Real-world Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: THALIA-01
Record Dates: First submitted 2022-02-07; First posted 2022-02-09 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational Group: Patients receive TKIs after T-DM1 progression.
  Interventions: Drug: TKIs

INTERVENTIONS:
Drug: TKIs — tyrosine kinase inhibitors based therapy

SUMMARY:
This is a real world study to evaluate the efficacy and safety of tyrosine kinase inhibitors after T-DM1 progression.

DETAILED DESCRIPTION:
HER2-positive breast cancers account for 15%-20% of all breast cancers. The development of HER2 targeted therapies have greatly improved the survival of HER2-positive breast cancer patients. Trastuzumab emtansine (T-DM1) has shown great effectiveness in treating HER2-positive metastatic breast cancer, but therapies subsequent to T-DM1 progression are still controversial. Here, we investigated efficacy and safety of tyrosine kinase inhibitors (TKIs) based therapy in T-DM1 resistant HER2-positive metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female and 18-70 years old
* Metastatic or locally recurrent HER2-positive breast cancer
* Patients received TKIs-based therapy after T-DM1 failure in treatment for metastasis
* Complete and accurate medical data

Exclusion Criteria:

- Incomplete medical data

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HER2-positive metastatic breast cancer patients who failed by T-DM1 received TKIs
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | 2 years
  Progression-free survival estimated using Kaplan-Meier methods is defined as the time from the date of informed consent to the earlier of death or disease progression. Patients alive without disease progression are censored at the date of last disease evaluation. Progressive disease (PD) based on RECIST 1.1 is at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Equivocal progression of non-target lesions also qualifies as PD.
Objective Response Rate (ORR) | 2 years
  The overall response rate is defined as the percentage of patients with a best overall response of CR or PR relative to the appropriate analysis set

SECONDARY OUTCOMES:
The Number of Participants Who Experienced Adverse Events (AE) | 2 years
  Safety will be assessed by standard clinical and laboratory tests (haematology, serum chemistry). AE grade were defined by the NCI CTCAE (National Cancer Institute Common Terminology Criteria for Adverse Events).

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Provincial People's Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No